CLINICAL TRIAL: NCT00538317
Title: Comparison of Administration of Tirofiban in the Ambulance or in the Cathlab in Patients With Acute Myocardial Infarction Treated With Primary Angioplasty
Brief Title: GPIIbIIIa Inhibitors in the RESCUe and RESURCOR Networks at the Acute Myocardial Infarction
Acronym: AGIR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Eric BONNEFOY-CUDRAZ, MD, Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-452
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction,; GPIIbIIIa inhibitors,; primary angioplasty,; tirofiban
MeSH Terms: interventions — Tirofiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): tirofiban bolus + perfusion started at the site of caring
  Interventions: Drug: tirofiban
- 2 (Active Comparator): tirofiban bolus + perfusion started at the beginning of coronarography (usual use of tirofiban)
  Interventions: Drug: tirofiban

INTERVENTIONS:
Drug: tirofiban — bolus of 25 µg/kg lasting 3 minutes then 18h to 24h perfusion of 0.15 µg/kg/min
  Other Names: agrastat
  Arms: 1
Drug: tirofiban — bolus of 25 µg/kg lasting 3 minutes then 18h to 24h perfusion of 0.15 µg/kg/min
  Other Names: agrastat
  Arms: 2

SUMMARY:
In patients with acute myocardial infarction who are managed in the prehospital setting, and who will treated with primary angioplasty, we evaluate the benefit of an early administration of tirofiban, a powerful GPIIbIIIa inhibitors. Patients are randomised to early administration in the ambulance or administration in the cathlab. The primary endpoint is TIMI 2-3 flow in the first coronary opacification of the culprit artery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Information given to the patient and consent obtained
* Thoracic pain or symptoms of infarction
* Symptoms < 12 hours
* ST deviation identified by electrocardiography (ECG) in at least 2 contiguous leads
* Transfer time to angioplasty room evaluated by the coordinating doctor as less than 90 minutes (from ECG diagnosis to arrival in angioplasty room)

Exclusion criteria

* Physiological or pathological conditions not compatible with a revascularisation procedure (in the acute phase of myocardial infarction (MI)
* Administration of fibrinolytics or another antiGPIIBIIIa in the previous seven days
* Contraindications to aspirin or tirofiban or heparin
* Diagnosed severe kidney failure (dialysis, creatinin > 350µmol/l
* Pregnancy
* Time for transfer to the angioplasty room evaluated by coordinating doctor as more than 90 minutes
* Subject participating in another trial
* Subject with high hemorrhagic risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
TIMI 2-3 flow on first coronary artery opacification | start of coronarography

SECONDARY OUTCOMES:
Protocol déviations of Tirofiban administration (no bolus, bolus decreasing or increasing of +/- 10% from expected value, dose perfusion decreasing or increasing of 1 ml/h from expected value, time perfusion > 24h or < 18h | During tirofiban administration
TIMI 3, TIMI 2 and TIMI 1-0 flow frequency in responsible artery before and after angioplasty | before and after angioplasty
left ventricular ejection fraction value | during angioplasty
CPK and troponin values (before and after angioplasty, peak and 24h after angioplasty) | during 24h after angioplasty
reduction of ST segment elevation (considered as resoluted if amplitude decreasing > 70%) | after angioplasty
Outcome of following Serious Adverse Events: anginal recurrence, infarct recurrence, urgent revascularization, serious heart failure and hospital mortality | During hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bonnefoy-Cudraz, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] El Khoury C, Dubien PY, Mercier C, Belle L, Debaty G, Capel O, Perret T, Savary D, Serre P, Bonnefoy E; AGIR-2 Investigators. Prehospital high-dose tirofiban in patients undergoing primary percutaneous intervention. The AGIR-2 study. Arch Cardiovasc Dis. 2010 May;103(5):285-92. doi: 10.1016/j.acvd.2010.04.005. Epub 2010 Jun 17. PMID 20619238